CLINICAL TRIAL: NCT05657327
Title: Application and Optimization of the International Study Group of Pancreatic Surgery (ISGPS) Definition and Grading Criteria for Postoperative Complications of Pancreatic Surgery in Laparoscopic Pancreatic Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xinrui Zhu，MD, Director, West China Hospital
Other Study IDs: 126059
Record Dates: First submitted 2022-12-10; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Laparoscopic Pancreatic Surgery; Pancreatic Fistula; Postoperative Bleeding; Delayed Gastric Emptying
MeSH Terms: conditions — Pancreatic Fistula; Postoperative Hemorrhage; Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with postoperative complications: Postoperative complications such as pancreatic fistula, postoperative bleeding and delayed gastric emptying
- Group without postoperative complications: No postoperative complications such as pancreatic fistula, postoperative bleeding and delayed gastric emptying

SUMMARY:
In recent years, with the continuous development of minimally invasive techniques, laparoscopic pancreatic surgery has also been widely used. Although the postoperative mortality rate of laparoscopic pancreatic surgery has been decreasing as the technology continues to improve and mature, the complication rate reported varies widely among centers.The definition and grading criteria of ISGPS on postoperative complications of pancreatic surgery are mostly proposed based on open pancreatic surgery, and most of the data of the later related studies are also for open pancreatic surgery, while the applicability of the definition and grading criteria in laparoscopic pancreatic surgery is still lacking in systematic The study The main purpose of this study is to investigate the applicability of the ISGPS definition and grading criteria for pancreatic fistula, postoperative bleeding and delayed gastric emptying in laparoscopic pancreatic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. All patients underwent laparoscopic pancreatic resections at the Department of Pancreatic Surgery of West China Hospital of Sichuan University and the Department of Minimal Invasive Surgery of Shangjin Nanfu Hospital between January 2014 and July 2022.
2. All patients underwent laparoscopic pancreaticoduodenectomy (LPD), laparoscopic distal pancreatectomy (LDP), laparoscopic enucleation, laparoscopic middle pancreatectomy (LMP), laparoscopic duodenum-preserving resection of head of pancreas (LDPRHP), or laparoscopic Frey procedure.
3. Patients whose demographic parameters, perioperative clinical variables, postoperative follow-up outcomes for 3 months and total hospital costs can be collected completely.

Exclusion Criteria:

1. Patients converted to laparotomy
2. Patients underwent total pancreatectomy
3. Patients underwent pancreatic pseudocyst drainage management
4. Patients underwent pancreas biopsy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. All patients underwent laparoscopic pancreatic resections at the Department of Pancreatic Surgery of West China Hospital of Sichuan University and the Department of Minimal Invasive Surgery of Shangjin Nanfu Hospital between January 2014 and July 2022.
  2. All patients underwent laparoscopic pancreaticoduodenectomy (LPD), laparoscopic distal pancreatectomy (LDP), laparoscopic enucleation, laparoscopic middle pancreatectomy (LMP), laparoscopic duodenum-preserving resection of head of pancreas (LDPRHP), or laparoscopic Frey procedure.
  3. Patients whose demographic parameters, perioperative clinical variables, postoperative follow-up outcomes for 3 months and total hospital costs can be collected completely.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Length of hospitalization | Entire perioperative period
  Including the patient's perioperative hospital stay, postoperative time to discharge, and length of stay in the ICU
Medical expenses | Entire perioperative period
  Including the entire hospitalization period, medicine, surgery, etc.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Result] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Result] Bassi C, Butturini G, Molinari E, Mascetta G, Salvia R, Falconi M, Gumbs A, Pederzoli P. Pancreatic fistula rate after pancreatic resection. The importance of definitions. Dig Surg. 2004;21(1):54-9. doi: 10.1159/000075943. Epub 2003 Dec 30. PMID 14707394
- [Result] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Result] Pratt WB, Maithel SK, Vanounou T, Huang ZS, Callery MP, Vollmer CM Jr. Clinical and economic validation of the International Study Group of Pancreatic Fistula (ISGPF) classification scheme. Ann Surg. 2007 Mar;245(3):443-51. doi: 10.1097/01.sla.0000251708.70219.d2. PMID 17435552
- [Result] Hackert T, Hinz U, Pausch T, Fesenbeck I, Strobel O, Schneider L, Fritz S, Buchler MW. Postoperative pancreatic fistula: We need to redefine grades B and C. Surgery. 2016 Mar;159(3):872-7. doi: 10.1016/j.surg.2015.09.014. Epub 2015 Oct 23. PMID 26603847
- [Result] Hassenpflug M, Hinz U, Strobel O, Volpert J, Knebel P, Diener MK, Doerr-Harim C, Werner J, Hackert T, Buchler MW. Teres Ligament Patch Reduces Relevant Morbidity After Distal Pancreatectomy (the DISCOVER Randomized Controlled Trial). Ann Surg. 2016 Nov;264(5):723-730. doi: 10.1097/SLA.0000000000001913. PMID 27455155
- [Result] Maggino L, Malleo G, Bassi C, Allegrini V, McMillan MT, Borin A, Chen B, Drebin JA, Ecker BL, Fraker DL, Lee MK, Paiella S, Roses RE, Salvia R, Vollmer CM Jr. Decoding Grade B Pancreatic Fistula: A Clinical and Economical Analysis and Subclassification Proposal. Ann Surg. 2019 Jun;269(6):1146-1153. doi: 10.1097/SLA.0000000000002673. PMID 31082914
- [Result] Wente MN, Veit JA, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Yeo CJ, Buchler MW. Postpancreatectomy hemorrhage (PPH): an International Study Group of Pancreatic Surgery (ISGPS) definition. Surgery. 2007 Jul;142(1):20-5. doi: 10.1016/j.surg.2007.02.001. PMID 17629996
- [Result] Wente MN, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Traverso LW, Yeo CJ, Buchler MW. Delayed gastric emptying (DGE) after pancreatic surgery: a suggested definition by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2007 Nov;142(5):761-8. doi: 10.1016/j.surg.2007.05.005. PMID 17981197
- [Result] Pulvirenti A, Marchegiani G, Pea A, Allegrini V, Esposito A, Casetti L, Landoni L, Malleo G, Salvia R, Bassi C. Clinical Implications of the 2016 International Study Group on Pancreatic Surgery Definition and Grading of Postoperative Pancreatic Fistula on 775 Consecutive Pancreatic Resections. Ann Surg. 2018 Dec;268(6):1069-1075. doi: 10.1097/SLA.0000000000002362. PMID 28678062